CLINICAL TRIAL: NCT04836377
Title: A Long-Term Follow-up Study of Subjects With Gaucher Disease Who Previously Received AVR-RD-02
Status: Terminated | Type: Observational
Why Stopped: This study was voluntarily terminated due to a business decision not to proceed, and not due to any safety or efficacy issue
Sponsor: AVROBIO (Industry)
Responsible Party: Sponsor
Other Study IDs: AVRO-RD-02-LTF01
Record Dates: First submitted 2021-03-23; First posted 2021-04-08 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2022-09

CONDITIONS: Type 1 Gaucher Disease
Keywords: Gaucher; Guard1
MeSH Terms: conditions — Gaucher Disease | interventions — Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood sample collections consisting of serum chemistry (and electrolytes), hematology, and urinalysis
  * Blood sample collection to assess for the presence of anti-GCase antibodies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with Gaucher 1 Disease: This is a long-term follow-up study of subjects who previously received AVR-RD-02 (single dose administration) in a preceding treatment study. No investigational product will be administered in this study.
  Interventions: Other: Safety and efficacy assessments

INTERVENTIONS:
Other: Safety and efficacy assessments — Safety evaluations, disease-specific assessments, and other assessments to monitor for long-term complications of gene therapy intervention
  Other Names: Gene Therapy Intervention

SUMMARY:
This is a multicenter, multinational long-term follow-up study to assess the long-term safety and durability of effect of AVR-RD-02 treatment in subjects who previously received AVR-RD-02 treatment (single dose administration).

DETAILED DESCRIPTION:
Subjects who received AVR-RD-02 in the preceding treatment study and who meet all eligibility criteria may participate in the AVRO-RD-02-LTF01 study. For individual participating subjects, the Baseline visit for the AVRO-RD-02-LTF01 study will coincide with the subject's last visit in the preceding treatment study, whenever feasible. Subjects will be asked to return for study visits at approximately 6-month intervals for the first 4 years of the study and then annually thereafter for 10 years (for a total follow-up of 14 years in this study), during which time periodic safety and efficacy assessments will be performed to assess measures of safety, engraftment, and clinical response after AVR-RD-02 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have been enrolled and received AVR-RD-02 as single dose administration
* Subject must be willing and able to provide written informed consent for the AVRO-RD-02-LTF01 study in accordance with applicable regulations and guidelines and to comply with all study visits and procedures.

Exclusion Criteria:

* Subject is currently enrolled in an AVROBIO-sponsored AVR-RD-02 treatment study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To permit longitudinal assessment of safety, efficacy and durability of effect of AVR-RD-02 gene therapy infusion in the AVRO-RD-02-LTF01 study, subjects must have received AVR-RD-02 in a preceding treatment study and agree to comply with the study visit schedule and procedures for AVRO-RD-02-LTF01 for inclusion in the Long-Term Follow-Up study.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline over time in spleen volume as assessed by abdominal Magnetic Resonance Imaging (MRI) | Baseline to Year 15 post gene therapy infusion
Baseline over time in liver volume as assessed by abdominal MRI | Baseline to Year 15 post gene therapy infusion
Baseline over time in hemoglobin | Baseline to Year 15 post gene therapy infusion
Change from Baseline over time in platelet count | Baseline to Year 15 post gene therapy infusion
Change from Baseline in plasma lyso-Gb1 levels by liquid chromatography tandem mass spectrometry (LC/MS/MS) | Baseline to Year 15 post gene therapy infusion
Incidence of newly-diagnosed malignancy, hematologic disorder, and/or immune related events/immunogenicity | Baseline to Year 15 post gene therapy infusion
Number of participants with clinically relevant abnormalities as assessed by vital signs | Baseline to Year 15 post gene therapy infusion
Number of participants with clinically relevant abnormalities, as assessed by physical examinations findings | Baseline to Year 15 post gene therapy infusion
Number of participants with clinically relevant abnormalities, as assessed by clinical laboratory tests | Baseline to Year 15 post gene therapy infusion
Number of participants with clinically relevant abnormalities, as assessed by electrocardiograms (ECGs) | Baseline to Year 15 post gene therapy infusion

SECONDARY OUTCOMES:
Change from baseline over time in glucocerebrosidase (GCase) GCase enzyme activity level in | Baseline to Year 15 post gene therapy infusion
Change from baseline over time in Enzyme Replacement Therapy (ERT) frequency and dosing | Baseline to Year 15 post gene therapy infusion
Changes in Gaucher biomarker indices of Gaucher disease in chitotriosidase enzyme activity levels in plasma | Baseline to Year 15 post gene therapy infusion
Changes in Gaucher biomarker indices of Gaucher disease in bone marrow burden (BMB) score as assessed by bone MRI | Baseline to Year 15 post gene therapy infusion
Changes in Gaucher biomarker indices of Gaucher disease in bone mineral density (BMD) as assessed by dual-energy X-ray absorptiometry (DXA) | Baseline to Year 15 post gene therapy infusion
Average Vector Copy Number (VCN) in bone marrow aspirate as assessed by quantitative polymerase chain reaction (qPCR) and/or droplet digital polymerase chain reaction (ddPCR) | Baseline to Year 15 post gene therapy infusion
Change from Baseline in anti-GCase total antibodies and subsequent titers by an electrochemiluminescence method | Baseline to Year 15 post gene therapy infusion
Changes in Gaucher disease in potential aberrant clonal expansion(s) assessed by performing insertional site analysis (ISA) | Baseline to Year 15 post gene therapy infusion
Presence of replication competent lentivirus (RCL) | Baseline to Year 15 post gene therapy infusion

CONTACTS AND LOCATIONS:
Overall Officials: Milena Veselinovic, MD, Study Director — AVROBIO
Locations (3):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Hackensack University Medical Center, Hackensack, New Jersey
- M.A.G.I.C. Clinic Ltd, Calgary, Calgary Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
To keep consistent with the current treatment listing